CLINICAL TRIAL: NCT03544970
Title: An Audit of the Posterior Fossa Characterization in Open Spina Bifida Based on Tertiary Center Experience
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s60814
Record Dates: First submitted 2018-05-17; First posted 2018-06-04 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Fetal Anomaly; Spinal Dysraphism; Chiari Malformation Type 2
Keywords: fetal MRI; Posterior fossa
MeSH Terms: conditions — Congenital Abnormalities; Spinal Dysraphism; Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain stem and posterior fossa measurements in spina bifida aperta fetuses to compare them with normal population. Additionally, Describe the difference between pre- and postoperative findings.

DETAILED DESCRIPTION:
Spina bifida aperta (SBA), often referred to as myelomeningocele (MMC) or myeloschisis, is a devastating yet non-lethal congenital malformation with complex physical and neurodevelopmental sequelae. Its prevalence is approximately 4.9 per 10,000 live births in Europe and 3.17 in the United States. SBA results in motor and sensory deficits, their extension being defined by the upper level of the anatomical defect. These range, as the level increases, from bladder, bowel and sexual dysfunction, to involvement of the lower and even upper extremities, and secondary orthopaedic disabilities. Despite improvements in prevention, diagnosis, and postnatal management, SBA remains a major source of morbidity and mortality throughout the world. Children with SBA almost invariably have an associated Chiari II hindbrain malformation (CM II) and ventriculomegaly. The Chiari II malformation is characterized by posterior fossa (PF) and brain stem abnormalities, with downward displacement and compression of the cerebellum and brain stem.

Geerdink demonstrated that morphometric measures reliably quantify the morphological distortions of Chiari II malformation on postnatal MR images. These included downward herniation of the cerebellum, displacement of pons, medulla and fourth ventricle, medullary kinking, abnormal fourth ventricle, tentorium and mesencephalic tectum. The mamillopontine distance (MPD) and the cerebellar width were the most sensitive and specific determinant of Chiari II. Some foetuses with SBA have ventriculomegaly and its degree is believed to be predictive for the need of postnatal shunting.

In 2011, the Management of Myelomeningocele Study (MOMS) demonstrated the benefit of in utero repair of MMC as the need for ventricular shunting at 12 months was reduced and motor outcome at 30 months improved. Fetuses with the suspicion of SBA should be assessed comprehensively to counsel parents about the expected outcome and whether they would be candidates for fetal surgery. In this assessment, fetal MR has a crucial role to characterize the extent of brain abnormalities, the level of the lesion, and to rule out additional anomalies in fetuses with SBA. For fetal surgery eligibility, the presence of CM II on MR is a necessary finding. Many measurements have been proposed to describe the typical PF changes in fetuses with SBA, yet the reproducibility of these has rarely been studied. These include the transverse cerebellar diameter (TCD), the transverse diameter of the posterior fossa (TDPF), the midsagittal PF area, the level of cerebellar herniation and the clivus-supraocciput angle (CSA). These parameters have also been shown to change after in utero repair of SBA in small series and at different time points after fetal surgery, yet no study has consistently reported early postoperative assessment in utero.

The aims of this study were threefold: (1) to assess the reproducibility of measurements of the brain stem and PF that have been suggested to be representative on postnatal 8,9 and prenatal MR imaging (2) apply those parameters that were shown to be reproducible, to discriminate fetuses with SBA from gestational age matched fetuses with a normal PF; (3) and document early changes in these measurements one week after fetal surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients were those having fetal MR examination for additional assessment because of the prenatal diagnosis of SBA on ultrasound.
* appropriate gestational age - matched controls. The latter were fetuses assessed for other congenital anomalies, which do not affect the central nervous system (CNS) or were scanned for suspected CNS abnormalities with normal prenatal US, fetal MR and normal postnatal evaluation

Exclusion Criteria:

* twin pregnancy, syndromal pathology, fetal hydrops or anhydramnios.
* poor image quality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant
Study Population: Fetuses with spina bifida aperta with an additiona lsubgroup of matched pairs with pre- and postoperative imaging
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
(1) assess the reliability of brain stem and posterior fossa measurements and compare the reliable ones with a normal populations (2) and between paired pre- and postsurgical fetuses | Examinations from 2011 - 2016
  Biometric variables include the transverse cerebellar diameter (TCD), Transverse diameter of the fossa posterior (TDPF), the midsagittal PF area. The ventricular width will be measured in the coronal plane according to Garel and in case of asymmetry the largest value will be taken into account. Mammilopontine distande (MPD), the level of kinking of the brain stem, medullary length, tentorial length and width of the cisterna magna will be measured. The width of the foramen magnum is defined as the distance between opisthion to the basion. Tonsillar level (TL) will be measured by drawing a perpendicular line from the foramen magnum to the lowest cerebellar portion. In the presence of cerebellar herniation the deepest portion will be used. The cerebellopontine angle will also be measured.
  These are all metric data and will be reported in mm. To adjust for normal changes according to gestational age, there will be a correction based on an observed/expeted ratio for the parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium